CLINICAL TRIAL: NCT02787460
Title: Testing the Effectiveness of Behavioral Text Messages to Promote Attendance at HMRE Sessions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mathematica Policy Research, Inc. (Other)
Collaborators: Department of Health and Human Services (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MPR-500098-UF
Record Dates: First submitted 2016-05-26; First posted 2016-06-01 (Estimated); Last update posted 2021-02-02 (Actual); Status verified 2021-01

CONDITIONS: Family Relations; Marriage
Keywords: Parenting; Family Relations; Marriage; Relationships

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Behavioral Text Messages (Experimental): Couples assigned to a treatment group will receive weekly behavioral theory-based messages encouraging them to attend the sessions.
  Interventions: Behavioral: Behavioral Text Messages
- Simple Reminder Text Messages (No Intervention): Couples in the control group will receive "simple" reminder text messages that include the date, time, and location of their next group session

INTERVENTIONS:
Behavioral: Behavioral Text Messages
  Arms: Behavioral Text Messages

SUMMARY:
The University of Florida offers relationship education programs named ELEVATE, for couples, and Smart Steps, for couples in stepfamilies, in Citrus, Duval, Manatee, Palm Beach, and Santa Rosa counties. Each workshop comprises 4 2.5-hour long sessions. The STREAMS evaluation will examine whether text messages informed by behavioral insight theory can improve couples' attendance at relationship skills education group sessions, and if so, which kinds of messages are most effective

DETAILED DESCRIPTION:
The University of Florida operates the SMART program, which will offer four relationship education programs, each targeting a different population: (1) Relationship Smarts PLUS, for high school youth; (2) Before You Tie the Knot, for couples interested in marriage; (3) ELEVATE, for couples, and (4) Smart Steps, for couples in stepfamilies. All programming is offered through the University of Florida's IFAS Extension service in Citrus, Duval, Manatee, Palm Beach, and Santa Rosa counties.

The STREAMS evaluation will test text messaging strategies with couples enrolled in ELEVATE and Smart Steps. It will examine whether text messages informed by behavioral insight theory can improve couples' attendance at relationship skills education group sessions, and if so, which kinds of messages are most effective. ACF staff have noted that among the most common technical assistance requests from HMRE grantees are help with improving participation. Even if relationship skills sessions are offered in a convenient location where adults receive other services and even if programs offer transportation, child care and other assistance to facilitate regular program attendance, achieving consistent participation in these voluntary programs can be challenging. The University of Florida study will help address these challenges by examining whether text messages based on behavioral theories can work as a simple, practical strategy for improving program participation in group sessions. More broadly, the site will also add to the large and growing effort across the federal government to study the use of behavioral interventions or "nudges" to improve social programs.

ELIGIBILITY:
Inclusion Criteria:

* Couple
* Both partners consent to receive text messages

Exclusion Criteria:

* Single Adults
* Either Partner or both do not consent to receive text messages

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1904 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2020-04 (Actual); Study Completion 2020-04 (Actual)

PRIMARY OUTCOMES:
Attendance at programming session | Within 1 month of baseline
  Whether couple attends all 4 group programming sessions

CONTACTS AND LOCATIONS:
Overall Officials: Diane Paulsell, Principal Investigator — Mathematica Policy Research
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No